CLINICAL TRIAL: NCT03611998
Title: Survivors of Sex Trafficking: Occupation-Based Interventions for Executive Functioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSUHSCIRB9383
Record Dates: First submitted 2018-07-02; First posted 2018-08-02 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Sex Trafficking; Mental Disorder
Keywords: Sex trafficking; Occupational therapy; Occupation-based programming; Activity-based programming; Brain trauma
MeSH Terms: conditions — Mental Disorders; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: One group, pretest-posttest design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Survivors of Sex Trafficking (Experimental): Survivors of sex trafficking (SST) who were living in a residential facility participated in this project by receiving occupation-based programming to address limitations in executive function skills over the course of the 8-month project. Sessions were held twice-monthly for an hour duration at each session.
  Interventions: Behavioral: Occupation-based programming

INTERVENTIONS:
Behavioral: Occupation-based programming — Group sessions consisted of specific tasks performed to completion that emphasized skills such as problem-solving, decision-making, frustration tolerance, appropriate pacing, attention, inquiring, sequencing, gathering, organizing, adjusting, responding, enduring, initiating and cooperating. Examples of tasks included projects that the women were specifically interested in learning such as jewelry making, holiday decorations, clay work and other home décor projects. Investigators observed these and other behaviors during the group sessions, and scored individuals using the OTTOS instrument.

SUMMARY:
Persons traumatized through sex trafficking can demonstrate similar neurobehavioral and executive function (EF) deficits as persons with cortical injuries. In this pilot study, occupation-based activity (OBA) programming was implemented at a residence for females who had been trafficked. The study hypothesis was that OBA would facilitate development of EF skills in these clients, enabling more successful occupational performance. Method: Eight women engaged in OBA sessions over the course of eight months. Session objectives were to maximize independence in daily life skills and to foster EF component skills such as problem-solving, decision-making, cooperation, direction following and appropriate self-expression. Outcome measures used were the Executive Function Performance Test (EFPT), the Canadian Occupational Performance Measure (COPM) and the Occupational Therapy Task Observation Scale (OTTOS). Results: Gains were seen from baseline to final session in COPM score changes meeting minimally clinical difference, and OTTOS scores showing significant improvement: t(7)= -2.49, p=.04. Preliminary findings suggest that occupation-based programming may facilitate development of EF skills in sex-trafficked women.

DETAILED DESCRIPTION:
Individuals who are sex-trafficked experience a combination of sexual violence, emotional trauma, and physical injuries that lead to high rates of depression, anxiety and post traumatic stress disorder (PTSD) Prolonged stress and adverse learning experiences can also cause use-dependent brain changes that influence executive functioning (EF) development. Other distressing situations, such as living in poverty or in dangerous environments and experiencing early sexual trauma, can result in interrupted development of executive functioning skills Although the current OT literature in the area of human and sex trafficking provide recommendations regarding areas of advocacy, education and occupation-based interventions, there is no empirical evidence to date investigating the efficacy of occupation-based interventions with survivors of sex trafficking (SST). The research question addressed in this pilot study was whether occupation-based interventions would improve the overall occupational performance of SST living in a residential program. Therefore, the purpose was to objectively determine the efficacy of occupation-based activity to improve EF skills in SST; the researchers expected that an improvement in EF skills would translate to improved occupational performance.

This pilot study used a one-group, pretest-posttest design. Participants in the study were residents of a local residential program for survivors of sex trafficking (SST). Eight women, average age, 20 to 50 years who were living in the home during the eight-month project period, engaged in the occupation-based intervention groups provided and completed assessment outcome measures (Canadian Occupational Performance Measure and the Executive Function Performance Test) before and after completing the program. Group behavior was scored at each session attended with the Occupational Therapy Task Observation Scale (OTTOS). Group sessions consisted of specific tasks performed to completion that emphasized problem-solving, decision-making, frustration tolerance and cooperation.

Current performance level rating and performance satisfaction scores from the COPM, as well as scores from each area of the EFPT, were collected upon initial evaluation and at the end of the eight-month intervention period. OTTOS scores were recorded during each group intervention for individual clients and graphically recorded to demonstrate individual changes over time; day one OTTOS scores were compared to the OTTOS score of the final intervention. All comparisons were completed using two-tailed, paired t-tests with a .05 alpha level for significance.

ELIGIBILITY:
Inclusion Criteria:

* Participant had to be a resident of the performance site and have a history of being sex-trafficked.

Exclusion Criteria:

* Participants were not enrolled if behavioral issues prevented participation or impacted the safety of others as determined by resident directors

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Project performance site was a residential facility for women who were sex-trafficked; Typically women are the gender involved in this activity.
Enrollment: 8 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Executive Function Performance Test (EFPT) | 8 months
  The EFPT is a task-based measure where clients engage in actual functional tasks, including a simple cooking activity, use of telephone to obtain public information, organization of a medication routine, and money management. The number of cues needed to perform each task and the type of cue used is recorded. The EFPT measures the construct of executive function.

SECONDARY OUTCOMES:
The Canadian Occupational Performance Measure (COPM) | 8 months
  The COPM measures the construct of occupational performance. The tool consists of an unstructured interview whereby the rater assists the client in articulating current daily activities in the domains of self-care, work, and leisure. From this list of activities, the client rates the importance of each activity and her current satisfaction with performance on each task. A prioritized list of the five most important activities is created and associated satisfaction levels are assigned. The list can serve as a foundation for intervention planning and creation of client-centered goals.
The Occupational Therapy Task Observation Scale (OTTOS) | 8 months
  The OTTOS evaluates task and general behavior. Skills subsumed under task behavior measured by the OTTOS include 1) engagement; 2)coordination, 3) follows directions, 4) quality of work, 5) independence, 6) initiative, 7) decision making, 8) concentration, 9) frustration tolerance, and 10) problem solving; skills subsumed under general behavior include 11) appearance, 12) activity level, 13) expression, 14) cooperation, and 7) socialization. Each skill is scored on a 10-point rating scale, 0 being dysfunctional, and 10 being functional. A total score for task behavior is generated (max 100) and a total score for general behavior is multiplied by 2, to also obtain a max of 100. The tool is frequently used with clients having psychiatric disorders and has shown a high correlation (0.92) between occupational therapist raters.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon W. Mangum, MPS, LOTR, Principal Investigator — Louisiana State University Health Sciences Center
Locations (1):
- Louisiana State University Health Sciences Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Babcock, E. (2014). Using brain science as a way out of poverty. Crittenton Women's Union. @http://s3.amazonaws.com/empath-website/pdf/Research-UsingBrainScienceDesignPathwaysPoverty-0114.pdf.
- [Background] Hemmings S, Jakobowitz S, Abas M, Bick D, Howard LM, Stanley N, Zimmerman C, Oram S. Responding to the health needs of survivors of human trafficking: a systematic review. BMC Health Serv Res. 2016 Jul 29;16:320. doi: 10.1186/s12913-016-1538-8. PMID 27473258
- [Background] Newby A, McGuinness TM. Human trafficking: what psychiatric nurses should know to help children and adolescents. J Psychosoc Nurs Ment Health Serv. 2012 Apr;50(4):21-4. doi: 10.3928/02793695-20120307-03. Epub 2012 Mar 14. PMID 22421012
- [Background] Perry, B. D. (2009). Examining child maltreatment through a neurodevelopmental lens: Clinical applications of the neurosequential model of therapeutics. Journal of Loss and Trauma, 14(4), 240-255. 10.1080/15325020903004350 Retrieved from https://doi.org/10.1080/15325020903004350
- [Background] Baum CM, Connor LT, Morrison T, Hahn M, Dromerick AW, Edwards DF. Reliability, validity, and clinical utility of the Executive Function Performance Test: a measure of executive function in a sample of people with stroke. Am J Occup Ther. 2008 Jul-Aug;62(4):446-55. doi: 10.5014/ajot.62.4.446. PMID 18712007
- [Background] Law M, Baptiste S, McColl M, Opzoomer A, Polatajko H, Pollock N. The Canadian occupational performance measure: an outcome measure for occupational therapy. Can J Occup Ther. 1990 Apr;57(2):82-7. doi: 10.1177/000841749005700207. PMID 10104738
- [Background] Margolis RL, Harrison SA, Robinson HJ, Jayaram G. Occupational therapy task observation scale (OTTOS): a rapid method for rating task group function of psychiatric patients. Am J Occup Ther. 1996 May;50(5):380-5. doi: 10.5014/ajot.50.5.380. PMID 8728668